CLINICAL TRIAL: NCT00763815
Title: A Randomized, Double-blind, Placebo-controlled, 2-arm Parallel-group, Multicenter Study With a 24-week Main Treatment Period and an Extension Assessing the Efficacy and Safety of AVE0010 on Top of Pioglitazone in Patients With Type 2 Diabetes Not Adequately Controlled With Pioglitazone
Brief Title: GLP-1 Receptor Agonist Lixisenatide in Patients With Type 2 Diabetes for Glycemic Control and Safety Evaluation, on Top of Pioglitazone
Acronym: GETGOAL-P
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC6017; EudraCT: 2007-005884-92
Record Dates: First submitted 2008-09-30; First posted 2008-10-01 (Estimated); Results first posted 2016-10-11 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes Mellitus Type 2
Keywords: hyperglycemia GLP-1 pioglitazone
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — lixisenatide; Pioglitazone; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lixisenatide (Experimental): 2-step initiation regimen of lixisenatide: 10 microgram (mcg) once daily (QD) for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to the end of treatment.
  Interventions: Drug: Lixisenatide (AVE0010); Device: Pen auto-injector; Drug: Pioglitazone; Drug: Metformin
- Placebo (Placebo Comparator): 2-step initiation regimen of volume matching placebo: 10 mcg QD for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to the end of treatment.
  Interventions: Drug: Placebo; Device: Pen auto-injector; Drug: Pioglitazone; Drug: Metformin

INTERVENTIONS:
Drug: Lixisenatide (AVE0010) — Self-administered by subcutaneous injections once daily within the hour preceding breakfast.
  Arms: Lixisenatide
Drug: Placebo — Self-administered by subcutaneous injections once daily within the hour preceding breakfast.
  Arms: Placebo
Device: Pen auto-injector
  Other Names: OptiClik®
Drug: Pioglitazone — Dose to be kept stable.
Drug: Metformin — Metformin, if given to be continued at stable dose (at least 1.5 gram per day) up to the end of treatment.

SUMMARY:
The purpose of this study is to evaluate the benefits and risks of lixisenatide (AVE0010), in comparison to placebo, as an add-on treatment to pioglitazone with or without metformin, over a period of 24 weeks of treatment, followed by an extension.

The primary objective is to assess the effects of lixisenatide when added to pioglitazone on glycemic control in terms of glycosylated hemoglobin (HbA1c) reduction (absolute change) at Week 24.

Secondary objectives are to assess the effects of lixisenatide when added to pioglitazone on the percentage of patients reaching HbA1c less than 7 percent (%) and less than or equal to 6.5%, fasting plasma glucose (FPG), body weight, beta-cell function (assessed by homeostatic model assessment of beta-cell function [HOMA-beta]), and on fasting plasma insulin (FPI), to assess the safety, tolerability, pharmacokinetics (PK) and anti-lixisenatide antibody development.

DETAILED DESCRIPTION:
Patients who complete the 24-week main double-blind treatment would undergo a variable double-blind extension treatment, which ends for all patients at approximately the schedule date of Week 76 visit (Visit 25) for the last randomized patients.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus, diagnosed for at least 1 year at the time of the screening visit, insufficiently controlled with pioglitazone

Exclusion Criteria:

* HbA1c less than (<) 7 percent (%) or greater than (>) 10% at screening
* At the time of screening age <legal age of majority
* Pregnant or breastfeeding women and women of childbearing potential without effective contraceptive method of birth control
* Type 1 diabetes mellitus
* Pioglitazone not at a stable dose of at least 30 milligram per day (mg/day) for at least 3 months prior to screening
* If treatment with metformin, no stable dose of at least 1.5 gram per day (g/day) for at least 3 months prior to screening visit
* FPG at screening >250 milligram per deciliter (mg/dL) (>13.9 millimole per liter [mmol/L])
* Body mass index less than or equal to (<=) 20 kilogram per square meter (kg/m^2)
* Weight change of more than 5 kg during the 3 months preceding the screening visit
* History of unexplained pancreatitis, chronic pancreatitis, pancreatectomy, stomach/gastric surgery, or inflammatory bowel disease
* History of metabolic acidosis, including diabetic ketoacidosis within 1 year prior to screening
* Hemoglobinopathy or hemolytic anemia, or receipt of blood or plasma products within3 months prior to the time of screening
* History of myocardial infarction or stroke within the last 6 months prior to screening
* Known history of drug or alcohol abuse within 6 months prior to the time of screening
* Cardiovascular, hepatic, neurological, endocrine disease, active malignant tumor or other major systemic disease or patients with short life expectancy making implementation of the protocol or interpretation of the study results difficult, history or presence of clinically significant diabetic retinopathy, history or presence of macular edema likely to require laser treatment within the study period
* Uncontrolled or inadequately controlled hypertension at the time of screening with a resting systolic blood pressure or diastolic blood pressure (DBP) >180 millimeter of mercury (mmHg) or >95 mmHg, respectively
* Laboratory findings at the time of screening: aspartate aminotransferase (AST), alanine aminotransferase (ALT), or alkaline phosphatase (ALP): >2 times upper limit of normal (ULN) laboratory range; amylase and/or lipase: >3 times ULN; total bilirubin: >1.5 times ULN (except in case of Gilbert's syndrome); Hemoglobin <11 gram/deciliter and/or neutrophils <1500 per cubic millimeter (mm^3) and/or platelets <100 000/mm^3; positive test for Hepatitis B surface antigen (HBsAg) and/or Hepatitis C antibody (HCAb); positive serum pregnancy test in females of childbearing potential
* Any clinically significant abnormality identified on physical examination, laboratory tests, electrocardiogram (ECG), or vital signs at the time of screening that, in the judgment of the investigator or any sub-investigator, precludes safe completion of the study or constrains efficacy assessment
* Patients who are considered by the investigator or any sub-investigator as inappropriate for this study for any reason (for example, impossibility to meet specific protocol requirements [such as scheduled visits, being able to do self-injections]; likelihood of requiring treatment during the screening phase and treatment phase with drugs not permitted by the clinical study protocol; investigator or any sub-investigator, pharmacist, study coordinator, other study staff or relative thereof directly involved in the conduct of the protocol)
* Use of other oral or injectable antidiabetic or hypoglycemic agents other than metformin or pioglitazone (for example, sulfonylurea, alpha-glucosidase inhibitor, other thiazolidinediones, rimonabant, exenatide, dipeptidyl peptidase-4 [DPP-4] inhibitors, insulin) within 3 months prior to the time of screening
* Use of systemic glucocorticoids (excluding topical application or inhaled forms) for 1 week or more within 3 months prior to the time of screening
* Use of any investigational drug within 3 months prior to study
* Any previous treatment with lixisenatide or participation in a previous study with lixisenatide
* Renal impairment defined with creatinine >1.4 mg/dL in women and creatinine >1.5 mg/dL in men (applicable only for patients with metformin treatment)
* Patients with cardiac failure or history of cardiac failure (New York Heart Association class I to IV)
* End-stage renal disease defined by a serum creatinine clearance of <15 milliliter per minute (mL/min) (calculated by the Cockcroft and Gault formula) and/or patients on dialysis, if no treatment with metformin
* Clinically relevant history of gastrointestinal disease associated with prolonged nausea and vomiting, including, but not limited to, gastroparesis and gastroesophageal reflux disease requiring medical treatment, within 6 months prior to the time of screening
* Allergic reaction to any glucagon like peptide-1 (GLP-1) agonist in the past (for example,exenatide, liraglutide) or to metacresol
* Additional exclusion criteria at the end of the run-in phase: informed consent withdrawal; lack of compliance during the single-blind placebo run-in phase (>2 injections missed); and patient with any adverse event which precludes the inclusion in the study, as assessed by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 484 (Actual)
Dates: Start 2008-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (150):
- United States (85):
  - Sanofi-Aventis Investigational Site Number 840723, Birmingham, Alabama
  - Sanofi-Aventis Investigational Site Number 840744, Birmingham, Alabama
  - Sanofi-Aventis Investigational Site Number 840867, Birmingham, Alabama
  - Sanofi-Aventis Investigational Site Number 840720, Birmingham, Alabama
  - Sanofi-Aventis Investigational Site Number 840855, Mobile, Alabama
  - Sanofi-Aventis Investigational Site Number 840863, Mobile, Alabama
  - Sanofi-Aventis Investigational Site Number 840775, Chandler, Arizona
  - Sanofi-Aventis Investigational Site Number 840722, Mesa, Arizona
  - Sanofi-Aventis Investigational Site Number 840769, Phoenix, Arizona
  - Sanofi-Aventis Investigational Site Number 840729, Harrisburg, Arkansas
  - Sanofi-Aventis Investigational Site Number 840776, Mountain Home, Arkansas
  - Sanofi-Aventis Investigational Site Number 840795, Artesia, California
  - Sanofi-Aventis Investigational Site Number 840782, Chino, California
  - Sanofi-Aventis Investigational Site Number 840785, Huntington Beach, California
  - Sanofi-Aventis Investigational Site Number 840858, La Jolla, California
  - Sanofi-Aventis Investigational Site Number 840784, Los Banos, California
  - Sanofi-Aventis Investigational Site Number 840773, Mission Hills, California
  - Sanofi-Aventis Investigational Site Number 840707, Mission Viejo, California
  - Sanofi-Aventis Investigational Site Number 840733, Northridge, California
  - Sanofi-Aventis Investigational Site Number 840864, Roseville, California
  - Sanofi-Aventis Investigational Site Number 840772, San Diego, California
  - Sanofi-Aventis Investigational Site Number 840743, San Mateo, California
  - Sanofi-Aventis Investigational Site Number 840721, Stockton, California
  - Sanofi-Aventis Investigational Site Number 840763, West Hills, California
  - Sanofi-Aventis Investigational Site Number 840872, Colorado Springs, Colorado
  - Sanofi-Aventis Investigational Site Number 840868, Colorado Springs, Colorado
  - Sanofi-Aventis Investigational Site Number 840727, Jacksonville, Florida
  - Sanofi-Aventis Investigational Site Number 840745, New Port Richey, Florida
  - Sanofi-Aventis Investigational Site Number 840761, Oviedo, Florida
  - Sanofi-Aventis Investigational Site Number 840799, Wellington, Florida
  - Sanofi-Aventis Investigational Site Number 840857, Augusta, Georgia
  - Sanofi-Aventis Investigational Site Number 840724, Idaho Falls, Idaho
  - Sanofi-Aventis Investigational Site Number 840791, Chicago, Illinois
  - Sanofi-Aventis Investigational Site Number 840738, Avon, Indiana
  - Sanofi-Aventis Investigational Site Number 840794, Indianapolis, Indiana
  - Sanofi-Aventis Investigational Site Number 840767, Kansas City, Kansas
  - Sanofi-Aventis Investigational Site Number 840779, Lansing, Kansas
  - Sanofi-Aventis Investigational Site Number 840739, Wichita, Kansas
  - Sanofi-Aventis Investigational Site Number 840789, Lexington, Kentucky
  - Sanofi-Aventis Investigational Site Number 840850, Lexington, Kentucky
  - Sanofi-Aventis Investigational Site Number 840862, Baton Rouge, Louisiana
  - Sanofi-Aventis Investigational Site Number 840879, Shreveport, Louisiana
  - Sanofi-Aventis Investigational Site Number 840764, Hyattsville, Maryland
  - Sanofi-Aventis Investigational Site Number 840871, Rockville, Maryland
  - Sanofi-Aventis Investigational Site Number 840851, Russells Mills, Massachusetts
  - Sanofi-Aventis Investigational Site Number 840708, Kalamazoo, Michigan
  - Sanofi-Aventis Investigational Site Number 840774, Bloomington, Minnesota
  - Sanofi-Aventis Investigational Site Number 840704, Eagan, Minnesota
  - Sanofi-Aventis Investigational Site Number 840717, Picayune, Mississippi
  - Sanofi-Aventis Investigational Site Number 840765, St Louis, Missouri
  - Sanofi-Aventis Investigational Site Number 840875, Las Vegas, Nevada
  - Sanofi-Aventis Investigational Site Number 840866, Pahrump, Nevada
  - Sanofi-Aventis Investigational Site Number 840865, New York, New York
  - Sanofi-Aventis Investigational Site Number 840766, New York, New York
  - Sanofi-Aventis Investigational Site Number 840874, Staten Island, New York
  - Sanofi-Aventis Investigational Site Number 840762, West Seneca, New York
  - Sanofi-Aventis Investigational Site Number 840747, Burlington, North Carolina
  - Sanofi-Aventis Investigational Site Number 840760, Greensboro, North Carolina
  - Sanofi-Aventis Investigational Site Number 840712, High Point, North Carolina
  - Sanofi-Aventis Investigational Site Number 840780, Bismarck, North Dakota
  - Sanofi-Aventis Investigational Site Number 840877, Fargo, North Dakota
  - Sanofi-Aventis Investigational Site Number 840777, Athens, Ohio
  - Sanofi-Aventis Investigational Site Number 840741, Cleveland, Ohio
  - Sanofi-Aventis Investigational Site Number 840728, Dayton, Ohio
  - Sanofi-Aventis Investigational Site Number 840709, Mentor, Ohio
  - Sanofi-Aventis Investigational Site Number 840716, Norman, Oklahoma
  - Sanofi-Aventis Investigational Site Number 840701, Medford, Oregon
  - Sanofi-Aventis Investigational Site Number 840751, Beaver, Pennsylvania
  - Sanofi-Aventis Investigational Site Number 840798, Red Lion, Pennsylvania
  - Sanofi-Aventis Investigational Site Number 840792, Columbia, South Carolina
  - Sanofi-Aventis Investigational Site Number 840740, Simpsonville, South Carolina
  - Sanofi-Aventis Investigational Site Number 840726, Taylors, South Carolina
  - Sanofi-Aventis Investigational Site Number 840711, Bristol, Tennessee
  - Sanofi-Aventis Investigational Site Number 840853, Colleyville, Texas
  - Sanofi-Aventis Investigational Site Number 840730, Houston, Texas
  - Sanofi-Aventis Investigational Site Number 840854, San Antonio, Texas
  - Sanofi-Aventis Investigational Site Number 840796, Clinton, Utah
  - Sanofi-Aventis Investigational Site Number 840755, Salt Lake City, Utah
  - Sanofi-Aventis Investigational Site Number 840756, Salt Lake City, Utah
  - Sanofi-Aventis Investigational Site Number 840758, Salt Lake City, Utah
  - Sanofi-Aventis Investigational Site Number 840753, Norfolk, Virginia
  - Sanofi-Aventis Investigational Site Number 840770, Norfolk, Virginia
  - Sanofi-Aventis Investigational Site Number 840752, Richmond, Virginia
  - Sanofi-Aventis Investigational Site Number 840757, Virginia Beach, Virginia
  - Sanofi-Aventis Investigational Site Number 840735, Spokane, Washington
- Austria (6):
  - Sanofi-Aventis Investigational Site Number 040706, Graz
  - Sanofi-Aventis Investigational Site Number 040702, Vienna
  - Sanofi-Aventis Investigational Site Number 040704, Vienna
  - Sanofi-Aventis Investigational Site Number 040701, Vienna
  - Sanofi-Aventis Investigational Site Number 040705, Vienna
  - Sanofi-Aventis Investigational Site Number 040707, Wels
- Canada (10):
  - Sanofi-Aventis Investigational Site Number 124716, Greater Sudbury
  - Sanofi-Aventis Investigational Site Number 124710, London
  - Sanofi-Aventis Investigational Site Number 124712, Mirabel
  - Sanofi-Aventis Investigational Site Number 124705, Saint Romuald
  - Sanofi-Aventis Investigational Site Number 124703, Saskatoon
  - Sanofi-Aventis Investigational Site Number 124713, Scarborough
  - Sanofi-Aventis Investigational Site Number 124711, Sherbrooke
  - Sanofi-Aventis Investigational Site Number 124704, Smiths Falls
  - Sanofi-Aventis Investigational Site Number 124701, Thornhill
  - Sanofi-Aventis Investigational Site Number 124708, Vancouver
- France (5):
  - Sanofi-Aventis Investigational Site Number 250704, Armentières
  - Sanofi-Aventis Investigational Site Number 250707, La Rochelle
  - Sanofi-Aventis Investigational Site Number 250705, Labarthe-sur-Lèze
  - Sanofi-Aventis Investigational Site Number 250702, Le Creusot
  - Sanofi-Aventis Investigational Site Number 250701, Strasbourg
- Germany (7):
  - Sanofi-Aventis Investigational Site Number 276708, Aßlar
  - Sanofi-Aventis Investigational Site Number 276704, Berlin
  - Sanofi-Aventis Investigational Site Number 276703, Künzing
  - Sanofi-Aventis Investigational Site Number 276706, Leipzig
  - Sanofi-Aventis Investigational Site Number 276707, Pirna
  - Sanofi-Aventis Investigational Site Number 276702, Sulzbach-Rosenberg
  - Sanofi-Aventis Investigational Site Number 276701, Würzburg
- Greece (4):
  - Sanofi-Aventis Investigational Site Number 300705, Athens
  - Sanofi-Aventis Investigational Site Number 300703, Athens
  - Sanofi-Aventis Investigational Site Number 300704, Athens
  - Sanofi-Aventis Investigational Site Number 300701, Thessaloniki
- Guatemala (4):
  - Sanofi-Aventis Investigational Site Number 320702, Guatemala City
  - Sanofi-Aventis Investigational Site Number 320701, Guatemala City
  - Sanofi-Aventis Investigational Site Number 320703, Guatemala City
  - Sanofi-Aventis Investigational Site Number 320704, Guatemala City
- India (4):
  - Sanofi-Aventis Investigational Site Number 356701, Bangalore
  - Sanofi-Aventis Investigational Site Number 356703, Bangalore
  - Sanofi-Aventis Investigational Site Number 356702, Hyderabad
  - Sanofi-Aventis Investigational Site Number 356704, Nagpur
- Mexico (3):
  - Sanofi-Aventis Investigational Site Number 484703, Mérida
  - Sanofi-Aventis Investigational Site Number 484701, Tlalnepantla
  - Sanofi-Aventis Investigational Site Number 484704, Zapopan
- Peru (4):
  - Sanofi-Aventis Investigational Site Number 604703, Lima
  - Sanofi-Aventis Investigational Site Number 604701, Lima
  - Sanofi-Aventis Investigational Site Number 604702, Lima
  - Sanofi-Aventis Investigational Site Number 604705, Lima
- Puerto Rico (2):
  - Sanofi-Aventis Investigational Site Number 630714, Carolina
  - Sanofi-Aventis Investigational Site Number 630715, Carolina
- Romania (14):
  - Sanofi-Aventis Investigational Site Number 642711, Alba Iulia
  - Sanofi-Aventis Investigational Site Number 642702, Bacau
  - Sanofi-Aventis Investigational Site Number 642709, Baia Mare
  - Sanofi-Aventis Investigational Site Number 642701, Brasov
  - Sanofi-Aventis Investigational Site Number 642712, Bucharest
  - Sanofi-Aventis Investigational Site Number 642714, Bucharest
  - Sanofi-Aventis Investigational Site Number 642705, Constanța
  - Sanofi-Aventis Investigational Site Number 642707, Galati
  - Sanofi-Aventis Investigational Site Number 642703, Ploieşti
  - Sanofi-Aventis Investigational Site Number 642713, Reşiţa
  - Sanofi-Aventis Investigational Site Number 642708, Satu Mare
  - Sanofi-Aventis Investigational Site Number 642706, Târgu Mureş
  - Sanofi-Aventis Investigational Site Number 642715, Timișoara
  - Sanofi-Aventis Investigational Site Number 642710, Timișoara
- Turkey (Türkiye) (2):
  - Sanofi-Aventis Investigational Site Number 792702, Erzurum
  - Sanofi-Aventis Investigational Site Number 792705, Istanbul

REFERENCES:
- [Result] Pinget M, Goldenberg R, Niemoeller E, Muehlen-Bartmer I, Guo H, Aronson R. Efficacy and safety of lixisenatide once daily versus placebo in type 2 diabetes insufficiently controlled on pioglitazone (GetGoal-P). Diabetes Obes Metab. 2013 Nov;15(11):1000-7. doi: 10.1111/dom.12121. Epub 2013 May 26. PMID 23627775

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 150 centers in 13 countries between September 29, 2008 and June 29, 2011. The overall duration of treatment was at least 76 weeks (24 weeks main double-blind treatment; variable double-blind extension treatment).
Pre-assignment Details: A total of 906 patients were screened of which 422 (46.6%) were screen failures; main reason for screen failure was glycosylated hemoglobin (HbA1c) values being out of the defined protocol range (greater than or equal to 7% and less than or equal to 10%). A total of 484 patients were randomized.
Groups:
- Placebo: 2-step initiation regimen of volume matching placebo: 10 microgram (mcg) once daily (QD) subcutaneously for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to the end of treatment.
- Lixisenatide: 2-step initiation regimen of lixisenatide: 10 mcg QD subcutaneously for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to the end of treatment.
Period: Overall Study
Arm/Group | Placebo | Lixisenatide
Started | 161 (Randomized.) | 323
Treated/Safety Population | 161 (All patients who were exposed to at least 1 dose, regardless of amount of treatment administered.) | 323
Modified Intent-to-Treat(mITT)Population | 159 (All patients who received at least 1 dose;had baseline,at least 1 post-baseline efficacy assessment.) | 320
Completed | 109 | 239
Not Completed | 52 | 84
Not completed — Adverse Event | 14 | 29
Not completed — Lack of Efficacy | 10 | 11
Not completed — Poor Compliance to Protocol | 6 | 6
Not completed — Lost to Follow-up | 2 | 4
Not completed — Early Termination | 1 | 0
Not completed — Familial and Personal Reasons | 9 | 16
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 7 | 12
Not completed — Protocol Violation | 2 | 5
Not completed — Sponsor's Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized patients who were exposed to at least 1 dose of study drug, regardless of the amount of treatment administered.
Groups:
- Placebo: 2-step initiation regimen of volume matching placebo: 10 mcg QD subcutaneously for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to the end of treatment.
- Lixisenatide: 2-step initiation regimen of lixisenatide: 10 mcg once daily QD subcutaneously for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to the end of treatment.
- Total: Total of all reporting groups
Arm/Group | Placebo | Lixisenatide | Total
Number analyzed (Participants) | 161 | 323 | 484
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (9.5) | 56.0 (9.5) | 55.8 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 151 | 230
  Male | 82 | 172 | 254
Race/Ethnicity, Customized [Number; unit: participants]
  Race: Caucasian/White | 132 | 273 | 405
  Race: Black | 9 | 14 | 23
  Race: Asian/Oriental | 8 | 14 | 22
  Race: Other | 12 | 22 | 34
  Ethnicity: Hispanic | 41 | 87 | 128
  Ethnicity: Non Hispanic | 120 | 236 | 356
Glycosylated Hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of hemoglobin] | 8.06 (0.79) | 8.08 (0.90) | 8.07 (0.86)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: millimole per liter (mmol/L)] | 9.13 (2.20) | 9.11 (2.15) | 9.12 (2.16)
Body Weight [Mean (Standard Deviation); unit: kilogram] | 96.74 (25.58) | 92.93 (22.90) | 94.20 (23.87)
Beta-cell Function Assessed by Homeostasis Model Assessment for Beta-cell Function (HOMA-beta) [Mean (Standard Deviation); unit: percentage of normal beta cells function] — Beta cell function was assessed by HOMA-beta. HOMA-beta (% of normal beta cells function) = (20 multiplied by fasting plasma insulin [micro unit per milliliter]) divided by (fasting plasma glucose [mmol/L] minus 3.5). Here, Number of patients analyzed = 141 and 300 for Placebo and Lixisenatide treatment arms, respectively.
  percentage of normal beta cells function | 36.23 (26.50) | 34.69 (30.30) | 35.18 (29.12)
Fasting Plasma Insulin (FPI) [Mean (Standard Deviation); unit: picomole per liter (pmol/L)] — Here, Number of patients analyzed = 142 and 300 for Placebo and Lixisenatide treatment arms, respectively.
  picomole per liter (pmol/L) | 66.07 (48.12) | 63.32 (57.69) | 64.21 (54.76)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 8.09 (5.58) | 8.11 (5.44) | 8.10 (5.48)
Duration of Pioglitazone Treatment [Mean (Standard Deviation); unit: years] | 1.79 (2.51) | 1.69 (2.00) | 1.72 (2.18)
Pioglitazone Daily Dose [Number; unit: participants]
  >=30 milligram (mg) to Less Than (<) 45 mg | 126 | 242 | 368
  >= 45 mg | 35 | 81 | 116
Metformin Use at Screening [Number; unit: participants] — Number of patients with metformin use at baseline was reported.
  participants | 131 | 261 | 392
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] — BMI was calculated by dividing body weight (kilogram) by the height (meter) squared.
  kilogram per square meter (kg/m^2) | 34.44 (7.04) | 33.66 (6.71) | 33.92 (6.82)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 24
Description: Absolute change = HbA1c value at Week 24 minus HbA1c value at baseline. The on-treatment period for this efficacy variable is time from the first dose of study drug and up to 3 days after the last dose of study drug, on or before Visit 12 (Week 24) or Day 169 if Visit 12 is not available, and before the introduction of rescue therapy. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: mITT population:all randomized patients who received at least 1 dose;had baseline,at least 1 post-baseline efficacy assessment, irrespective of compliance with study protocol/procedures. Last observation carried forward used. Number of patients analyzed=patients with baseline and at least 1 post-baseline HbA1c assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: percentage of hemoglobin
Groups:
- Placebo: 2-step initiation regimen of volume matching placebo.
- Lixisenatide: 2-step initiation regimen of lixisenatide.
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 148 | 308
percentage of hemoglobin | -0.34 (0.100) | -0.90 (0.089)
Statistical Analysis 1: Comparison: Placebo vs Lixisenatide; To detect a difference of 0.5% (or 0.4%) in change from baseline to Week 24 in HbA1c between lixisenatide and placebo, 300 patients in lixisenatide arm and 150 patients in placebo arm would provide a power of 96% (or 86%) assuming common standard deviation of 1.3% with a 2-sided test at 5% significance level; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistical testing: 2-sided at significance level=0.05. Analysis of co-variance (ANCOVA) included treatment arms; randomization strata of screening HbA1c (<8.0, >=8.0%), metformin use (yes, no); country as fixed effects; baseline HbA1c as covariate; Least Squares (LS) Mean Difference = -0.56, 95% CI 2-sided [-0.731 to -0.386], Standard Error of Mean 0.088

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24
Description: Change was calculated by subtracting baseline value from Week 24 value. The on-treatment period for this efficacy variable is time from the first dose of study drug and up to 1 day after the last dose of study drug, on or before Visit 12 (Week 24) or Day 169 if Visit 12 is not available, and before the introduction of rescue therapy. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: mITT population. Missing data was imputed using last observation carried forward (LOCF). Here, number of patients analyzed = patients with baseline and at least 1 post-baseline FPG assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 159 | 317
mmol/L | -0.32 (0.215) | -1.16 (0.192)

3. Secondary Outcome: Change From Baseline in Body Weight at Week 24
Description: Change was calculated by subtracting baseline value from Week 24 value. The on-treatment period for this efficacy variable is time from the first dose of study drug and up to 3 days after the last dose of study drug, on or before Visit 12 (Week 24) or Day 169 if Visit 12 is not available, and before the introduction of rescue therapy. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: mITT population. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline body weight assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: kilogram
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 157 | 315
kilogram | 0.21 (0.357) | -0.21 (0.324)

4. Secondary Outcome: Change From Baseline in Fasting Plasma Insulin (FPI) at Week 24
Description: as for outcome 2
Time Frame: Baseline, Week 24
Population: mITT population. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline FPI assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 125 | 281
pmol/L | -1.01 (4.080) | -10.36 (3.397)

5. Secondary Outcome: Percentage of Patients With Glycosylated Hemoglobin (HbA1c) Level Less Than 7% at Week 24
Description: The on-treatment period for this efficacy variable is the time from the first dose of study drug up to 3 days after the last dose of study drug or up to the introduction of rescue therapy, whichever is the earliest. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Week 24
Population: mITT population. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline HbA1c assessment during on-treatment period.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 148 | 308
percentage of participants | 26.4 | 52.3

6. Secondary Outcome: Percentage of Patients With HbA1c Level Less Than or Equal to 6.5% at Week 24
Description: as for outcome 5
Time Frame: Week 24
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 148 | 308
percentage of participants | 10.1 | 28.9

7. Secondary Outcome: Change From Baseline in Beta-cell Function Assessed by Homeostasis Model Assessment for Beta-cell Function (HOMA-beta) at Week 24
Description: Beta cell function was assessed by HOMA-beta. HOMA-beta (% of normal beta cells function) = (20 multiplied by fasting plasma insulin [micro unit per milliliter]) divided by (fasting plasma glucose [mmol/L] minus 3.5). Change was calculated by subtracting baseline value from Week 24 value. The on-treatment period for this efficacy variable is time from the first dose of study drug and up to 1 day after the last dose of study drug, on or before Visit 12 (Week 24) or Day 169 if Visit 12 is not available, and before the introduction of rescue therapy. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: mITT population. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline HOMA-beta assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: % of normal beta cells function
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 124 | 281
% of normal beta cells function | 6.98 (3.575) | 6.72 (2.963)

8. Secondary Outcome: Percentage of Patients Requiring Rescue Therapy During Main 24-Week Period
Description: Routine fasting self-monitored plasma glucose (SMPG) and central laboratory FPG (and HbA1c after week 12) values were used to determine the requirement of rescue medication. If fasting SMPG value exceeded the specified limit for 3 consecutive days, the central laboratory FPG (and HbA1c after week 12) were performed. Threshold values - from baseline to Week 8: fasting SMPG/FPG >270 milligram/deciliter (mg/dL) (15.0 mmol/L), from Week 8 to Week 12: fasting SMPG/FPG >240 mg/dL (13.3 mmol/L), and from Week 12 to Week 24: fasting SMPG/FPG >200 mg/dL (11.1 mmol/L) or HbA1c >8.5%. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline up to Week 24
Population: mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 159 | 320
percentage of participants | 11.3 | 3.8

9. Other Pre Specified Outcome: Percentage of Patients With at Least 5% Weight Loss From Baseline at Week 24
Description: The on-treatment period for this efficacy variable is time from the first dose of study drug and up to 3 days after the last dose of study drug, on or before Visit 12 (Week 24) or Day 169 if Visit 12 is not available, and before the introduction of rescue therapy. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: mITT population. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline body weight assessment during on-treatment period.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 157 | 315
percentage of participants | 5.1 | 9.2

10. Other Pre Specified Outcome: Number of Patients With Symptomatic Hypoglycemia and Severe Symptomatic Hypoglycemia
Description: Symptomatic hypoglycemia was an event with clinical symptoms that were considered to result from a hypoglycemic episode with an accompanying plasma glucose less than 60 mg/dL (3.3 mmol/L) or associated with prompt recovery after oral carbohydrate, intravenous glucose, or glucagon administration if no plasma glucose measurement was available. Severe symptomatic hypoglycemia was symptomatic hypoglycemia event in which the patient required the assistance of another person and was associated with either a plasma glucose level below 36 mg/dL (2.0 mmol/L) or prompt recovery after oral carbohydrate, intravenous glucose, or glucagon administration, if no plasma glucose measurement was available.
Time Frame: First dose of study drug up to 3 days after the last dose administration, for up to 132 weeks
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 161 | 323
participants
  Symptomatic Hypoglycemia | 7 | 23
  Severe Symptomatic Hypoglycemia | 0 | 0

ADVERSE EVENTS:
Time Frame: First dose of study drug up to 3 days after the last dose administration, for up to 132 weeks
Description: Median exposure to study treatment was 615.5 and 588.0 days in lixisenatide and placebo treatment arms, respectively. The analysis was performed on safety population, defined as all randomized patients who were exposed to at least 1 dose of study drug, regardless of the amount of treatment administered.
Arm/Group | Placebo | Lixisenatide
Serious Adverse Events (participants affected / at risk) | 15/161 | 25/323
Other Adverse Events (participants affected / at risk) | 105/161 | 219/323
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=161) | Lixisenatide (N=323)
Appendicitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 1 | 0
Diabetic foot infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Memory impairment (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Diabetic retinopathy (Eye disorders) | 0 | 1
Macular oedema (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1
Vitreous haemorrhage (Eye disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 1
Mitral valve incompetence (Cardiac disorders) | 1 | 0
Blue toe syndrome (Vascular disorders) | 0 | 1
Shock haemorrhagic (Vascular disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 2
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Stag horn calculus (Renal and urinary disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 3
Blood calcitonin increased (Investigations) | 1 | 0
Colonoscopy (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Abdominal injury (Injury, poisoning and procedural complications) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1
Coronary angioplasty (Surgical and medical procedures) | 0 | 1
Coronary artery bypass (Surgical and medical procedures) | 2 | 0
Percutaneous coronary intervention (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=161) | Lixisenatide (N=323)
Bronchitis (Infections and infestations) | 16 | 25
Influenza (Infections and infestations) | 9 | 24
Nasopharyngitis (Infections and infestations) | 24 | 53
Upper respiratory tract infection (Infections and infestations) | 18 | 41
Urinary tract infection (Infections and infestations) | 11 | 24
Hypoglycaemia (Metabolism and nutrition disorders) | 8 | 25 — Hypoglycaemia adverse event is based on investigator reported hypoglycaemia.
Dizziness (Nervous system disorders) | 13 | 33
Headache (Nervous system disorders) | 19 | 43
Hypertension (Vascular disorders) | 9 | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 18
Diarrhoea (Gastrointestinal disorders) | 23 | 35
Nausea (Gastrointestinal disorders) | 22 | 84
Vomiting (Gastrointestinal disorders) | 8 | 26
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 24
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 22
Fatigue (General disorders) | 3 | 21
Oedema peripheral (General disorders) | 9 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.